CLINICAL TRIAL: NCT05602896
Title: Reducing 30-Day Sepsis Readmissions: Impact of a Post Discharge Education Program
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decided to table the study
Sponsor: Washington University School of Medicine (Other)
Collaborators: BJC HealthCare (Other); Viven Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202207066
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Sepsis
Keywords: sepsis; education; cancer
MeSH Terms: conditions — Sepsis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sepsis Education (Experimental): The patient will receive a daily notification via their mobile phone and conduct the daily activity for 30 days. The program is interactive and aimed at measures that prevent exposure to infection sources in the environment, as well as recognition of early signs of infection and possible sepsis. Each session takes approximately 2 minutes or less. Each scenario or session has the user identify where germs may be present and then asks the user to perform a simple action to remove the germs (e.g. with an antiseptic wipe). The range of activities include cleaning of surfaces, proper mask use, and hand sanitizing. This includes areas of their home such as the kitchen, bathroom, living room/family room. The program also addresses common community areas such as public transit, grocery stores, and restaurants
  Interventions: Other: Sepsis education

INTERVENTIONS:
Other: Sepsis education — The education program has been reviewed and approved by BJH Center for Practice Excellence

SUMMARY:
This study will advance the knowledge in the field by determining the effectiveness of discharge education regarding prevention of a new infection which is the highest cause of readmission for sepsis patient. In evaluating the impact care teams will develop a clearer link between specific home-based education interventions and infection prevention. This study is an exploratory study designed to identify whether patient education through an innovative teaching method can have an impact on readmissions. This study may the first of several based on findings from this initial, exploratory study.

ELIGIBILITY:
Inclusion Criteria:

* Oncology patients discharged to home following a diagnosis of sepsis, severe sepsis or septic shock
* Patient must have a mobile phone/device
* English speakers
* Age range 18 - 85 years

Exclusion Criteria:

* Less than 18 years of age and older than 85 years of age
* No mobile phone/device
* Non-English speaking
* No diagnosis of sepsis, severe sepsis, or septic shock
* Non-Oncology patient

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-31 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Readmission rates | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Bickel, MSN, APRN, ANCP-BC, ACNS-BC, Principal Investigator — BJC HealthCare

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu